CLINICAL TRIAL: NCT05003440
Title: Investigation of Safety, Tolerability and Pharmacokinetic Properties of Multiple Doses of Oral NNC0385-0434 in Healthy, Male Japanese Participants
Brief Title: A Research Study Looking at How the Medicine NNC0385-0434 Works in the Body of Healthy Japanese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6435-4748; U1111-1264-4546 (Other: World Health Organization (WHO)); jRCT2071210055 (Registry Identifier: JAPIC)
Record Dates: First submitted 2021-08-10; First posted 2021-08-12 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers; Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Intervention Model Description: The study consists of two parts. Part 1 consists of three sequential dose ascension cohorts each with 4 healthy Japanese participants, randomised 3:1. The purpose of Part 1 is to provide safety clearance for initiating Part 2 and the randomisation of Japanese participants into the phase 2 study NN6435-4697. Part 2 will randomise the remaining Japanese participants into three parallel dose groups. (3:1:3:1:3:1).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- NNC0385-0434 15 mg (Experimental): 15 mg oral NNC0385-0434 will be administered once-daily over 10 consecutive days
  Interventions: Drug: NNC0385-0434
- Placebo (NNC0385-0434 15 mg) (Placebo Comparator): Oral placebo will be administered once-daily over 10 consecutive days
  Interventions: Drug: Placebo
- NNC0385-0434 40 mg (Experimental): 40 mg oral NNC0385-0434 will be administered once-daily over 10 consecutive days
  Interventions: Drug: NNC0385-0434
- Placebo (NNC0385-0434 40 mg) (Placebo Comparator): Oral placebo will be administered once-daily over 10 consecutive days
  Interventions: Drug: Placebo
- NNC0385-0434 100 mg (Experimental): 100 mg oral NNC0385-0434 will be administered once-daily over 10 consecutive days
  Interventions: Drug: NNC0385-0434
- Placebo (NNC0385-0434 100 mg) (Placebo Comparator): Oral placebo will be administered once-daily over 10 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC0385-0434 — Participants will get 1 tablet (oral use) of NNC0385-0434 per day for 10 days in either 15, 40 or 100 mg
  Arms: NNC0385-0434 100 mg; NNC0385-0434 15 mg; NNC0385-0434 40 mg
Drug: Placebo — Participants will get 1 tablet (oral use) of placebo per day for 10 days
  Arms: Placebo (NNC0385-0434 100 mg); Placebo (NNC0385-0434 15 mg); Placebo (NNC0385-0434 40 mg)

SUMMARY:
The aim of this study is to look at how the study medicine works in the body and how it is removed from the body.

We are testing the study medicine to make a medicine that can help people lower their cholesterol level.

Participants will either get

1. NNC0385-0434 (a potential new medicine) in one of three different doses: 15 mg, 40 mg, or 100 mg.
2. placebo (a dummy medicine which looks like the study medicine but without any medicine).

Which treatment participants get is decided by chance. NNC0385-0434 is a new medicine and has not been approved by the Health Authorities (Centre for Drug Evaluation).

Participants will get 1 tablet per day for 10 days. The tablet will be handed out by a study doctor or site staff at the clinic and the study will last between 62 and 98 days.

Participants will have 7 clinic visits. One of these visits will be a 13-day, 12-night stay (V2) and the rest will be 1-day visits (V1 and V3 to V7).

At all visits, except the information visit, participants will have blood drawn along with other clinical checks.

Participants will be asked about their health, medical history and habits including mental health.

ELIGIBILITY:
Inclusion Criteria:

* Body weight greater than or equal to 54.0 kg.
* Body mass index (BMI) between 20.0 and 34.9 kg/m^2 (both inclusive).

Exclusion Criteria:

* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator.
* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From pre-dose (day 1) until completion of the post-treatment period at follow-up (day 65)
  Count of events

SECONDARY OUTCOMES:
AUC0-24h,0434,Day10,; the area under the NNC0385-0434 plasma concentration-time curve from time 0 to 24 h after last dose of oral NNC0385-0434 | From last dose (day 10) 0 to 24 hours post treatment (day 11)
  h*nmol/L
Cmax,0434,Day10,; the maximum plasma concentration of NNC0385-0434 after last dose of oral NNC0385-0434 | From last dose (day 10) 0 hours to post treatment follow-up (day 65)
  nmol/L
tmax,0434,Day10; the time to maximum observed plasma concentration of NNC0385-0434 after last dose of oral NNC0385-0434 | From last dose (day 10) 0 hours to post treatment follow-up (day 65)
  hours
t½,0434,Day10; the terminal half-life of NNC0385-0434 after last dose of oral NNC0385-0434 | From last dose (day 10) 0 hours to post treatment follow-up (day 65)
  hours
AUC0-24h,SNAC,Day10,; the area under the SNAC plasma concentration-time curve from time 0 to 24 h after last dose of oral NNC0385-0434 | From last dose (day 10) 0 to 24 hours post treatment (day 11)
  h*nmol/L
Cmax,SNAC,Day10; the maximum plasma concentration of SNAC after last dose of oral NNC0385-0434 | From last dose (day 10) 0 to 24 hours post treatment (day 11)
  nmol/L
tmax,SNAC,Day10; the time to maximum observed plasma concentration of SNAC after last dose of oral NNC0385-0434 | From last dose (day 10) 0 to 24 hours post treatment follow-up (day 11)
  hours
t½,SNAC,Day10; the terminal half-life of SNAC after last dose of oral NNC0385-0434 | From last dose (day 10) 0 to 24 hours post treatment follow-up (day 11)
  hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Hakata Clinic, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com